CLINICAL TRIAL: NCT07139717
Title: Evaluation of the Effectiveness of Stool Color Card in the Early Detection of Biliary Atresia: A Prospective Study.
Brief Title: Stool Card in Biliary Atresia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Hamed Ahmed, Principal Investigator, Assiut University
Other Study IDs: Stool card in biliary atresia
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stool Color Card; Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effectiveness of using a stool color card as a non-invasive screening tool for the early detection of biliary atresia, with the objective of improving early diagnosis rates and facilitating timely surgical intervention.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a rare but life-threatening liver disorder that affects infants, characterized by the progressive inflammation and fibrosis of the bile ducts, leading to biliary obstruction [1].

Early diagnosis and intervention are crucial - ideally before 60 days of age - as BA is a leading cause of liver transplantation in children if not diagnosed and treated promptly [2]. The traditional method of diagnosis involves the identification of clinical signs like jaundice and abnormal liver function tests, but this approach can delay the diagnosis, leading to irreversible liver damage. As a result, early detection is essential to improve outcomes and prevent the need for a liver transplant [3].

The stool color card (SCC) is a diagnostic tool that has gained significant attention in recent years as a non-invasive method for the early detection of biliary atresia [4]. Newborns with biliary atresia typically exhibit pale stools due to a lack of bile secretion [5].

The stool color card provides a simple way for parents or healthcare professionals to monitor changes in the stool color in newborns, providing an early indicator of potential biliary atresia [6,7]. The card features a range of colors that correspond to the different stages of stool color, allowing for easy comparison and identification of abnormal stool [8-11].

Despite the availability of SCCs, their effectiveness in routine screening programs remains understudied. There is a need to evaluate the utility of SCCs in improving early diagnosis rates of BA.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates and infants aged 1-90 days old.
2. Neonates and infants with direct (conjugated) hyperbilirubinemia (Conjugated hyperbilirubinemia is generally defined as a conjugated or direct bilirubin level greater than 1 mg/dL when the total bilirubin is less than 5 mg/dL or more than 20% of the total bilirubin if the total bilirubin is greater than 5 mg/dL) [12]
3. No contraindication for liver biopsy as considered the gold standard for diagnosis of biliary atresia e.g. coagulopathy.

Exclusion Criteria:

1 - Infants diagnosed with biliary atresia or other cholestatic liver diseases prior to enrollment.

2-Infants aged more than 90 days 3-Neonates and infants with indirect hyperbilirubinemia. 4-Those with contraindication to do liver biopsy

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of newborn infants screened using the stool color card during the first six months of life. Participants will be recruited from pediatric outpatient clinics and neonatal follow-up units, as well as infants admitted with suspected liver disease at [Name of Hospital/Region]. Both healthy infants and those later diagnosed with biliary atresia will be included to evaluate the diagnostic accuracy of the stool color card.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Stool Color Card in Early Detection of Biliary Atresia | First 3 months
  Diagnostic accuracy of the stool color card for early detection of biliary atresia (BA). Accuracy will be evaluated by sensitivity (proportion of BA cases detected), specificity (proportion of healthy infants correctly identified as not having BA), positive predictive value (PPV), and negative predictive value (NPV), compared to the reference standard of final diagnosis confirmed by imaging or surgery.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gu YH, Yokoyama K, Mizuta K, Tsuchioka T, Kudo T, Sasaki H, Nio M, Tang J, Ohkubo T, Matsui A. Stool color card screening for early detection of biliary atresia and long-term native liver survival: a 19-year cohort study in Japan. J Pediatr. 2015 Apr;166(4):897-902.e1. doi: 10.1016/j.jpeds.2014.12.063. Epub 2015 Feb 11. PMID 25681196
- [Background] Feldman AG, Sokol RJ. Neonatal Cholestasis. Neoreviews. 2013 Feb 1;14(2):10.1542/neo.14-2-e63. doi: 10.1542/neo.14-2-e63. PMID 24244109
- [Background] Madadi-Sanjani O, Kuebler JF, Uecker M, Pfister ED, Baumann U, Kunze-Hullmann B, Blaser J, Buck T, Petersen C. Province-Wide Stool Color Card Screening for Biliary Atresia in Lower-Saxony: Experiences with Passive Distribution Strategies and Results. Int J Neonatal Screen. 2021 Nov 4;7(4):75. doi: 10.3390/ijns7040075. PMID 34842600
- [Background] Alam R, Nahid KL, Faruk MO, Rasna EH, Rukunuzzaman M. Use of stool color card as screening tool for biliary atresia in resource-constraint country. Gastroenterol Hepatol Bed Bench. 2024;17(2):146-150. doi: 10.22037/ghfbb.v17i2.2931. PMID 38994513
- [Background] El-Shabrawi MH, Baroudy SR, Hassanin FS, Farag AE. A pilot study of the value of a stool color card as a diagnostic tool for extrahepatic biliary atresia at a single tertiary referral center in a low/middle income country. Arab J Gastroenterol. 2021 Mar;22(1):61-65. doi: 10.1016/j.ajg.2020.12.004. Epub 2021 Mar 2. PMID 33664005
- [Background] Schreiber RA, Harpavat S, Hulscher JBF, Wildhaber BE. Biliary Atresia in 2021: Epidemiology, Screening and Public Policy. J Clin Med. 2022 Feb 14;11(4):999. doi: 10.3390/jcm11040999. PMID 35207269
- [Background] Rabbani T, Guthery SL, Himes R, Shneider BL, Harpavat S. Newborn Screening for Biliary Atresia: a Review of Current Methods. Curr Gastroenterol Rep. 2021 Nov 24;23(12):28. doi: 10.1007/s11894-021-00825-2. PMID 34817690